CLINICAL TRIAL: NCT04034511
Title: Impact of Medically-tailored Meals on Health Care Outcomes and Costs Among Low-income Adults With Diabetes
Brief Title: Food and Education Effects on Diabetes Study
Acronym: FEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Moveable Feast (Unknown); Priority Partners MCO (Unknown); Leonard & Helen R. Stulman Charitable Foundation (Unknown); France-Merrick Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00200526
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: nutrition; medically-tailored meals
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Nutrition Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor and data-analyst will be masked to treatment assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medically-tailored meal delivery and medical nutrition therapy (Experimental): Participants assigned to this arm will receive home-delivered, medically-tailored meals for 3 months combined with monthly individual Medical Nutrition Therapy sessions for 6 months. Participants will also receive participants' usual case management services from participants' Medicaid insurance program.
  Interventions: Other: Medically-tailored meal delivery and medical nutrition therapy
- Usual care (No Intervention): Participants assigned to this arm of the study will receive usual care and case management services from participants' Medicaid insurance program.

INTERVENTIONS:
Other: Medically-tailored meal delivery and medical nutrition therapy — Home-delivered, medically-tailored meals for 3 months combined with monthly individual medical nutrition therapy sessions for 6 months
  Arms: Medically-tailored meal delivery and medical nutrition therapy

SUMMARY:
Low-income adults are disproportionately affected by diabetes, experiencing greater rates of diabetes, diabetes-related complications, and mortality. Dietary habits play an important role in achieving and maintaining glycemic control to improve health outcomes. However, low-income adults are less likely to adopt the necessary dietary changes to improve glycemic control largely due to poor access to care, limited knowledge and skills to facilitate lifestyle change, and financial and environmental constraints that limit access to healthy foods. Nutrition interventions that target key barriers to healthy dietary habits among low-income adults with diabetes may have a profound impact on improving glycemic control. The provision of home-delivered, medically-tailored meals in addition to individualized medical nutrition therapy is a promising approach to improve dietary habits in socially disadvantaged populations with diabetes. Evidence suggests the provision of medically tailored meals may be beneficial in improving health outcomes and health care costs among socially disadvantaged adults with chronic illnesses, however rigorous studies specifically exploring the benefits of meal provision and medical nutrition therapy among adults with type 2 diabetes are lacking. The investigators aim to conduct a randomized-controlled clinical trial examining the impact of medically-tailored meals and medical nutrition therapy on health-related outcomes and health care costs among low-income adults with type 2 diabetes.

DETAILED DESCRIPTION:
The investigators will recruit 100 individuals age 18 and over with uncontrolled diabetes (defined as a hemoglobin A1c (HbA1c) >8%) and enrolled in Priority Partners Medicaid insurance. Participants will be randomized to one of two groups: 1) 3 months of home-delivered, medically-tailored meals combined with monthly individual Medical Nutrition Therapy sessions for 6 months or 2) usual care. The investigators will follow participants for up to 12 months to assess for changes in hemoglobin A1c.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Diabetes with a hemoglobin A1c>8%
* Medicaid beneficiary
* Enrolled in Medicaid Insurance

Exclusion Criteria:

* Medical conditions that are indications for additional dietary requirements (e.g., advanced chronic kidney disease, end-stage renal disease, chronic wounds, or severe alcohol use disorder)
* Swallowing difficulties
* Food allergies
* Non-English speaking
* Language or hearing impairment
* Currently pregnant or breast feeding
* Does not have a refrigerator/freezer in the home to store meals
* Has plans to move out of the meal delivery service area in the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin A1c | Baseline, 6 months
  Change in hemoglobin A1c (percent)

SECONDARY OUTCOMES:
Change in Hemoglobin A1c | Baseline, 12 months
  Change in Hemoglobin A1c (percent)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne M Clark, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clark JM, Maw MTT, Pettway K, Chander G, Elias S, Zisow-McClean S, Maruthur NM, Greer RC. Impact of Medically Tailored Meals on Clinical Outcomes Among Low-Income Adults with Type 2 Diabetes: A Pilot Randomized Trial. J Gen Intern Med. 2025 Jun;40(8):1711-1719. doi: 10.1007/s11606-024-09248-x. Epub 2024 Dec 13. PMID 39672984
- See also: France-Merrick Foundation — https://france-merrickfdn.org/